CLINICAL TRIAL: NCT06687200
Title: Evaluation of the Interest of a "Neutral Pelvic Positioning" on the Quality of Bone Repositioning in Patients Receiving Pelvic Radiotherapy
Brief Title: Assessing the Ompact of Neutral Pelvic Positioning on Bone Repositioning Quality in Pelvic Radiotherapy Patients
Acronym: Pelvtilt-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pelvtilt-RT ET23-309
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Radiotherapy; Repositonning Pelvic; Neutral Pelvic Positioning
Keywords: Neutral pelvic positioning; Radiotherapy; Image-Guided Radiotherapy; Glutes bridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Setup with neutral pelvic positioning technique (Experimental): Setup with neutral pelvic positioning technique (from dosimetry onward and at each session) and daily IGRT (CBCT or MVCT Mega Voltage Computed Tomography).
  Interventions: Other: Setup with neutral pelvic positioning technique
- Control Arm: Standard setup (Active Comparator): Standard setup (from dosimetry onward and at each session) and daily IGRT (CBCT or MVCT).
  Interventions: Other: Standard setup

INTERVENTIONS:
Other: Setup with neutral pelvic positioning technique — Setup with neutral pelvic positioning technique (from dosimetry onward and at each session) and daily IGRT (CBCT or MVCT Mega Voltage Computed Tomography)
  Arms: Experimental Arm: Setup with neutral pelvic positioning technique
Other: Standard setup — Standard setup (from dosimetry onward and at each session) and daily IGRT (CBCT or MVCT)
  Arms: Control Arm: Standard setup

SUMMARY:
This study explores whether achieving a neutral pelvic position improves bone repositioning quality for patients undergoing pelvic radiotherapy. While Intensity-Modulated Radiotherapy (IMRT) and Image-Guided Radiotherapy (IGRT) have enhanced target volume precision and reduced side effects, effective patient positioning remains crucial. However, rotational adjustments are limited without a specialized robotic table. Current immobilization devices, customizable or not, show limited impact on positioning accuracy, with mixed results on the use of knee and foot supports. A pilot study identified significant rotational variation, and to address this, a "glute bridge" maneuver is proposed to ensure a neutral pelvic position. This randomized study will evaluate the impact of this maneuver on positioning quality when combined with immobilization and skin markers.

DETAILED DESCRIPTION:
Radiotherapy (RT) is an integral part of curative treatment for pelvic cancers. Intensity-Modulated Radiotherapy (IMRT) has demonstrated benefits in target volume (TV) coverage and sparing healthy tissues. IMRT achieves a highly conformal dose distribution, with steep dose gradients between the TVs and Organs at Risk (OARs). However, its effectiveness depends on the quality of patient repositioning, ensured through positioning imaging, immobilization devices, and skin markers. Image-Guided Radiotherapy (IGRT) involves using imaging systems to verify the correct positioning of the patient, TVs, and OARs. IGRT has shown substantial benefits in enhancing treatment precision and reducing side effects. Translational adjustments can be applied before treatment, but, except for TomoTherapy®, which can correct roll, other rotations (pitch and yaw) require a 6D robotic table, a technology that is not widely available and limited to 3°.

The immobilization systems available and used in RT departments vary widely, classified into customizable and non-customizable systems. Two publications have shown that using a customizable immobilization system does not improve bone repositioning in these patients. Two teams have compared non-customizable immobilizations consisting of a knee support alone or combined with a foot support. The team of Cartal et al. (2015) found no significant difference in translations. However, using a knee support alone significantly reduced rotations over 3°. Laaksomaa et al. found no difference in performance between the two setups.

A pilot study in our department with 32 patients and nearly 700 images revealed an RX rotation greater than 3° in 19% of the images on average, ranging from 0% to 75% of the positioning images affected by an RX rotation over 3°. These patients were positioned supine with a knee support according to Cartal et al. Data, with a headrest or arm support added if lomboaortic irradiation was needed. Accessories were indexed, and their positions marked during the planning CT for reproducibility across sessions, with skin markers as additional setup aids.

Physical therapists recommend a maneuver called the "glute bridge," where patients bend their legs and lift their pelvis three times before straightening their legs without voluntary movement. For the study, the legs will rest on a reproducibly positioned knee support. This maneuver ensures a neutral pelvic position for each patient, relieving contractures in the lumbopelvic region. The "neutral zone" or "balance point theory," as defined by physiology and biomechanics, describes a state that relieves contractures in the lumbopelvic region and ensures balanced baseline tension across muscle groups. The pelvis lift creates co-contraction of the hamstrings, quadriceps, abdominals, and lumbar spinal muscles, promoting this balance.

In this randomized study, we propose evaluating the benefit of a neutral pelvic positioning setup achieved by the patient, in addition to immobilization devices and skin markers, on the quality of bone repositioning.

ELIGIBILITY:
Inclusion Criteria:

I1. Female, aged ≥ 18 years; I2. Patient scheduled for intensity-modulated radiotherapy for pelvic cancer, with an irradiation field extending at least up to L5-S1 on an accelerator equipped with a 3D imaging system (CBCT or MVCT) with automatic registration; I3. Patient affiliated with a social security scheme or equivalent; I4. Dated and signed informed consent.

Exclusion Criteria:

E1. Patient unable or unwilling to lift the pelvis; E2. Patient with anal or vulvar carcinoma; E3. Patient with unstable spondylolisthesis; E4. Patient with an unhealed lumbar or pelvic fracture; E5. Patient with a recent muscle injury in the relevant muscle groups; E6. Patient with an ECOG performance status ≥ 2; E7. Pregnant or breastfeeding patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The rate of images with RX > 3° will be calculated for each patient as the number of sessions with a repositioning image where RX is > 3°, relative to the total number of sessions performed. | At to 3 months

SECONDARY OUTCOMES:
The median, mean, and standard deviation of rotations (RX, RY, and RZ) obtained from the positioning imaging; | At to 3 months
The median, mean, and standard deviation of translations (TX, TY, and TZ) obtained from the positioning imaging | At to 3 months
The calculation of the dose delivered to nodal CTVs and organs at risk, recalculated by simulating the actual rotations observed during treatment | At to 24 months
Gastrointestinal, urinary, and hematological toxicities graded according to NCI-CTCAE v5 | Up to 24 months
Systematic error estimation calculated using the Van Herk et al. formula | At to 24 months
Random error estimation calculated using the Van Herk et al. formula | At to 24 months
Estimation of nodal CTV-PTV margins calculated using the Van Herk et al. formula | At to 24 months
Evaluation of repositioning error in relation to L4, without applying rotations, will be obtained using the mean and standard deviation of measurements between the anterosuperior part of the L4 vertebral body on the reference image and on the daily image | At to 3 months
  For irradiations including lombo-aortic nodal areas only
Evaluation of the RX rotation discrepancy observed after registering the daily image to the reference image, comparing two regions of interest: one defined by L1-L5 and the other defined from the iliac crests to the ischial tuberosities | At to 24 months
  For irradiations including lombo-aortic nodal areas only

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie de Lorraine, Nancy
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest - Saint-Herblain, Saint-Herblain